CLINICAL TRIAL: NCT05887011
Title: National Multicentre Non-interventional Study to Assess CRT Patterns and Short-term Outcomes on Unresectable NSCLC and SCLC in Routine Practices in Russia
Brief Title: CRT( Chemo-Radiation Therapy) Patterns and Short-term Outcomes on Unresectable NSCLC and SCLC in Routine Practices in Russia
Acronym: PASSAT
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00026
Record Dates: First submitted 2023-04-21; First posted 2023-06-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Unresectable /Inoperable Locally Advanced (Stage II-III) NSCLC and Locally Advanced LS-SCLC (Stage I-III)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LA NSCLC: unresectable/inoperable (stage II-III) locally advanced Non-Small Cell Lung Cancer
- LS-SCLC: unresectable/inoperable Limited-stage small cell lung carcinoma (stage I-III)

SUMMARY:
This is a multi-center, non-interventional, study with the aim to access routine practice of diagnostic and treatment approaches in patients with NSCLC and SCLC in 50 largest oncology centers in Russian Federation. The data for all 2000 patients with LA NSCLC and LS-SCLC who receiving CRT will have been collected for 2 years from the primary medical records. Demographic and clinical characteristics of the patients, information of routine diagnostics procedures and treatment approaches for patients with unresectable LA NSCLC and LS-SCLC and the treatment results of the end of CRT will be collected. Information about any specific NSCLC or SCLC treatments following CRT (e.g., durvalumab) will not be collected in the study. Patients with NSCLC and SCLC meeting the inclusion criteria will be prospectively enrolled into the study. Study procedures will comply with all the local regulatory requirements regarding AE reporting (pharmacovigilance). Study design considers secondary data collection approach using existing patients' medical records, after patients' visits according to routine sites' practice. Data for visit (record) 1 will be collected at the start of CRT (concurrent or sequential), and data for visit (record) 2 will be collected after the last dose of RT and with CT control results available, but the time frame for this data collection is expected to be no later than 6 months after visit 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Provision of written informed consent
3. Patient received at least one RT dose under prescribed CRT (concurrent or sequential) for definitive treatment of locally advanced NSCLC (stage II-III, unresectable or inoperable NSCLC, including locoregional recurrence and patient's refusal to undergo surgery) or LS-SCLC based on local MDT decision
4. Patient is currently undergoing RT (preferably no more than 10 doses)

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 months
2. Confirmation that the subject was already included in this study before
3. Absence of written informed consent form
4. Data erroneously collected from subjects for which written consent is not available, will not be included in or will be deleted from the study database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 2000 patients who received chemoradiotherapy (cCRT or sCRT) for the treatment of locally advanced NSCLC and SCLC in 50 largest oncology centers in Russian Federation. The total enrolment period will take up to 2 years. Information about specific NSCLC or SCLC treatments following CRT (e.g., durvalumab) will not be collected in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical characteristics of the population. NSCLC stage by TNM classification (% of patients). Patient status - locoregional recurrence and inoperable. Histology type. % of patients with known PD-L1 status and EGFR mutation status. | Baseline
  * % of patients with each TNM stage
  * % of patient with locoregional recurrence and inoperable patients (including patient's refusal)
  * Median age at the start of CRTs, % male/female, % of patients with comorbidities (and % by comorbidity type by MedDRA SOC/PT), % on concomitant medications,
  * % of patients by ECOG category;
  * % of patients with each tumour histology type;
  * % of patients with known PD-L1 status (and of those - % positive);
  * % of patients with known EGFR mutation status (and of those % by mutation status).
    * of patients with SCLC from all patients with locally or locally advanced LC receiving CRT
    * of patients with each TNM stage among SCLC
    * of pts with locoregional recurrence and inoperable pts among SCLC (including pt's refusal Median age at the start of CRTs, % male/female, % of patients with comorbidities (and % by comorbidity type by MedDRA SOC/PT), % on concomitant medications among SCLC
    * of patients by ECOG category among SCLC

SECONDARY OUTCOMES:
Chemoradiotherapy (CRT) details | up to 6 month
  · % of induction chemotherapy,
The short-term effectiveness results of the initial CRT treatment administered to patients with recently first diagnosed LA NSCLC or LS-SCLC (% of patients with CR, PR, ORR, SD, PD, unevaluable for response) for cCRT and sCRT respectively | up to 6 month
  * % of patients with CR,
  * % of patients with PR,
  * % of patients with OR (ORR),
  * % of patients with SD,
  * % of patients with PD,
  * % of patients unevaluable for response
Patterns of routine diagnostics and treatment for patients with unresectable LA NSCLC or LS-SCLC | up to 6 month
  Frequency distribution of each diagnostic approach applied;
Patterns of routine diagnostics and treatment for patients with unresectable LA NSCLC or LS-SCLC | up to 6 month
  Median time between the date patient first came to oncology center and the date of examination (by each approach);
Patterns of routine diagnostics and treatment for patients with unresectable LA NSCLC or LS-SCLC | up to 6 month
  Median time between the date of examination and date of start of CRT (by each approach);
Patterns of routine diagnostics and treatment for patients with unresectable LA NSCLC or LS-SCLC | up to 6 month
  Frequency distribution of results by categories (for example, staging, size, location, etc.) for each approach.
Chemoradiotherapy (CRT) details: concurrent CRT vs sequential CRT | up to 6 month
  Frequency distribution of patients who receive concurrent or sequential CRT
Chemoradiotherapy (CRT) details: presence of interruptions | up to 6 month
  % of CRT interruptions
Chemoradiotherapy (CRT) details: number of interruptions | up to 6 month
  average number of interruptions per patients
Chemoradiotherapy (CRT) details: durations of interruptions | up to 6 month
  median interruption duration (days) (based on mean duration per patient)
Chemoradiotherapy (CRT) details:Reasons for RT interruptions and dose reductions/ withdrawals; | up to 6 month
  frequency distribution of reasons to interrupt or stop RT
Chemoradiotherapy (CRT) details:· RT: doses, fractionation, planning, selective and elective irradiation of lymph nodes | up to 6 month
  frequency distribution of the number of RT fractions received
Chemoradiotherapy (CRT) details:· Type of platinum-based chemotherapy used | up to 6 month
  Frequency distribution of number chemotherapy courses, of types of platinum chemotherapy used
Chemoradiotherapy (CRT) details: For sCRT: duration between ChT and RT | up to 6 month
  For sCRT: range and median number of chemotherapy courses, median days between chemotherapy and radiotherapy
Chemoradiotherapy (CRT) details | up to 6 month
  · For ChT: number of chemotherapy courses
Chemoradiotherapy (CRT) details for SCLC | Up to 6 months
  Frequency distribution of the number of RT and doses received per day (2x1,5 Gy or 1X2 or 3 Gy)

CONTACTS AND LOCATIONS:
Locations (40):
- Russia (40):
  - Research Site, Arkhangelsk
  - Research Site, Balashikha
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Khabarovsk
  - Research Site, Khanty-Mansiysk
  - Research Site, Kirov
  - Research Site, Kostroma
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novokuznetsk
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Perm
  - Research Site, Podolsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saransk
  - Research Site, Saratov
  - Research Site, Sochi
  - Research Site, Syktivkar
  - Research Site, Tula
  - Research Site, Tver'
  - Research Site, Ulyanovsk
  - Research Site, Vladivostok
  - Research Site, Vologda
  - Research Site, Yakutia
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
  - Research Site, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home